CLINICAL TRIAL: NCT02573935
Title: A Randomized Placebo-controlled Phase II Study of Clarithromycin or Placebo Combined With VCD Induction Therapy Prior to High-dose Melphalan With Stem Cell Support in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Clarithromycin in Multiple Myeloma Induction Therapy
Acronym: CLAIM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Suspected side effects to the combination of clarithromycin and VCD (bortezomib, cyclophosphamide and dexamethasone)
Sponsor: Henrik Gregersen (Other)
Collaborators: Danish Myeloma Study Group (Other)
Responsible Party: Sponsor-Investigator, Henrik Gregersen, Consultant, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMSG 03/14; 2014-002187-32 (EudraCT Number)
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Clarithromycin; Induction Chemotherapy; Transplantation, Autologous
MeSH Terms: conditions — Multiple Myeloma | interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clarithromycin (Experimental): Clarithromycin combined with VCD induction therapy
  Interventions: Drug: Clarithromycin; Drug: VCD induction therapy
- Placebo (Placebo Comparator): Placebo combined with VCD induction therapy
  Interventions: Drug: Placebo; Drug: VCD induction therapy

INTERVENTIONS:
Drug: Clarithromycin — p.o. clarithromycin 500 mg twice daily for 63 days
  Arms: Clarithromycin
Drug: Placebo — Placebo tablet twice daily for 63 days
  Arms: Placebo
Drug: VCD induction therapy — Three courses of VCD (sc bortezomib 1.3 mg/sqm days 1, 4, 8, 11, iv cyclophosphamide 500 mg/sqm on days 1 and 8, and p.o. dexamethasone 40 mg days 1, 2, 4, 5, 8, 9, 11, 12 in each 21-days course)

SUMMARY:
This study evaluates the potential synergic anti-myeloma activity of clarithromycin when combined with VCD induction therapy in patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
The survival in younger myeloma patients improved in the nineties with the introduction of high-dose melphalan with autologous stem cell support (HDT). However, all patients will eventually experience relapse after HDT and there is a need for improvement of the response after HDT. The choice of induction treatment before HDT affects the outcome after induction therapy as well as the outcome after HDT.

Clarithromycin is a macrolide antibiotic frequently utilized in the treatment of respiratory tract infections and is often used in patients with known hypersensitivity to beta-lactam antibiotic. Besides antibiotic activity, clarithromycin may exert immunomodulatory and anti-inflammatory effects. The toxicity profile of clarithromycin is favourable and the cost is very low.

Studies on cell lines have shown that clarithromycin attenuates autophagy in myeloma cells and a recent study has demonstrated that treatment with clarithromycin enhanced bortezomib-induced cytotoxicity in myeloma cells. Phase II studies without control groups have indicated that clarithromycin might enhance the effect of the thalidomide and lenalidomide. A case-matched analysis compared patients at one centre receiving clarithromycin, lenalidomide and dexamethasone with an equal number of patients at another centre receiving lenalidomide and dexamethasone. This study indicated a favourable effect of clarithromycin with a higher frequency of complete response, very-good-partial-response or better response and progression-free survival. However, there is a need for controlled studies to determine whether clarithromycin might enhance the effect of other myeloma agents.

This randomized placebo-controlled study will include 160 patients with newly diagnosed multiple myeloma eligible for HDT. The study evaluates the potential synergic anti-myeloma activity of clarithromycin when combined with VCD induction therapy in patients with newly diagnosed multiple myeloma, and is conducted by the Danish Myeloma Study Group (DMSG) at seven clinics in Denmark. The first patient was included in May 2015 and enrolment is expected to continue until October 2016. The study ends when the last included patient has been followed for two months after HDT.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma diagnosis according to IMWG criteria
* Treatment demanding disease
* High-dose melphalan with stem cell support scheduled as a part of the treatment
* Signed informed consent given prior to any study related activities
* Age > 18 years

Exclusion Criteria:

* Allogeneic transplantation scheduled as a part of the treatment
* Myeloma treatment prior to entry in the study, except radiotherapy, bisphosphonates/denosumab or corticosteroids for symptom control
* Concurrent disease making clarithromycin treatment unsuitable
* Positive pregnancy test (only applicable for women with childbearing potential)
* Known or suspected hypersensitivity or intolerance to clarithromycin
* Prolonged QT corrected (QTc) interval ( > 500 msec on screening ECG)
* Concurrent treatment with cabergoline, fluconazole, ketoconazole, pimozide, quetiapine, sirolimus, verapamil, tacrolimus, ergot alkaloid, simvastatin or other statins
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrolment, uncontrolled angina or known cardiac amyloidosis
* Severe renal dysfunction (estimated creatinine clearance <10 mL/min)
* Serious medical or psychiatric illness which, in the judgment of the investigator, would make the patient inappropriate for entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Comparison of number of participants with very good partial response or better response after three courses of VCD combined with clarithromycin or placebo | 10 weeks

SECONDARY OUTCOMES:
Comparison of number of participants with very good partial response or better response after HDT in patients treated with three courses of VCD combined with clarithromycin or placebo | Five months
Comparison of number of participants with sCR, CR, PR, PD or SD in the treatment groups after induction therapy and HDT, respectively | Five months
Comparison of frequency of infections in patients treated VCD combined with clarithromycin or placebo | 9 weeks
Comparison of number of stem cells harvested in patients treated with clarithromycin and placebo in combination with VCD | Three months
Neurotoxicity assessed by FACT/GOG-Ntx, Version 4.0 | Five months
Quality of life assessed by EORTC QLQ-MY20 | Five months
Quality of life assessed by EORTC QLQ-C30 | Five months
Comparison of adverse events in patients treated VCD combined with clarithromycin or placebo assessed by CTCAE v4.0 | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Gregersen, MD, Principal Investigator — Aalborg University Hospital
Locations (7):
- Denmark (7):
  - Department of Hematology, Aalborg University Hospital, Aalborg
  - Department of Hematology, Aarhus University Hospital, Aarhus
  - Department of Hematology, Rigshospitalet, Copenhagen
  - Department of Hematology, Herlev Hospital, Herlev
  - Department of Hematology, Odense University Hospital, Odense
  - Department of Hematology, Roskilde Hospital, Roskilde
  - Department of Hematology, Vejle Hospital, Vejle

REFERENCES:
- [Background] Gay F, Rajkumar SV, Coleman M, Kumar S, Mark T, Dispenzieri A, Pearse R, Gertz MA, Leonard J, Lacy MQ, Chen-Kiang S, Roy V, Jayabalan DS, Lust JA, Witzig TE, Fonseca R, Kyle RA, Greipp PR, Stewart AK, Niesvizky R. Clarithromycin (Biaxin)-lenalidomide-low-dose dexamethasone (BiRd) versus lenalidomide-low-dose dexamethasone (Rd) for newly diagnosed myeloma. Am J Hematol. 2010 Sep;85(9):664-9. doi: 10.1002/ajh.21777. PMID 20645430
- [Derived] Nielsen LK, Klausen TW, Jarden M, Frederiksen H, Vangsted AJ, Do T, Kristensen IB, Frolund UC, Andersen CL, Abildgaard N, Gregersen H. Clarithromycin added to bortezomib-cyclophosphamide-dexamethasone impairs health-related quality of life in multiple myeloma patients. Eur J Haematol. 2019 Jan;102(1):70-78. doi: 10.1111/ejh.13175. Epub 2018 Oct 29. PMID 30230047
- [Derived] Gregersen H, Do T, Kristensen IB, Frolund UC, Andersen NF, Nielsen LK, Andersen CL, Klausen TW, Vangsted AJ, Abildgaard N. A randomized placebo-controlled phase II study of clarithromycin or placebo combined with VCD induction therapy prior to high-dose melphalan with stem cell support in patients with newly diagnosed multiple myeloma. Exp Hematol Oncol. 2018 Aug 13;7:18. doi: 10.1186/s40164-018-0110-0. eCollection 2018. PMID 30123673